CLINICAL TRIAL: NCT01966198
Title: Estimation of Autonomic Nervous System Modulation by Pulse Plethysmographic Analysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ASST Fatebenefratelli Sacco (Other)
Responsible Party: Principal Investigator, Riccardo Colombo, MD, ASST Fatebenefratelli Sacco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 31082013
Record Dates: First submitted 2013-10-12; First posted 2013-10-21 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Autonomic Nervous System Modulation
Keywords: pulse plethysmography, autonomic nervous system, heart rate variability, baro-reflex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- all patients (Experimental): tilt
  Interventions: Other: Tilt test

INTERVENTIONS:
Other: Tilt test — The experiment protocol consists of a sequence of passive postural changes gained with a tilt table, each of them lasting 10 minutes. The sequence consists of: (i) baseline recording in supine position; (ii) tilt at 45 degrees angle; (iii) recovery period in supine position; (iv) tilt at 90 degrees angle and (v) recovery in supine position.

SUMMARY:
Novel pulse plethysmography-derived indexes has been proposed as a tool to measure autonomic nervous system modulation in anaesthetized and awake patients, but nowadays a physiologic validation is lacking. We aim to examine the effects of sympathetic stimulation on pulse plethysmographic amplitude (PPGA), autonomic nervous system state (ANSS) and autonomic nervous system state index (ANSSi).

DETAILED DESCRIPTION:
It has been supposed that indexes derived from pulse plethysmographic analysis -the autonomic nervous system state (ANSS) and ANSS index (ANSSi)- may be useful tools to measure the autonomic nervous system (ANS) activity but, to date, physiologic experimental evidences are lacking.

Traditionally,it is widely accepted that ANS modulation and the baro-reflex control can be non-invasively studied through heart rate variability (HRV) and systolic variability analyses.

The aim of this study is to assess if PPGA-derived indexes are able to detect changes of ANS system modulation directed to heart and vessels.

Changes in position of patients lead to changes in the balance of the ANS. One of the most used manoeuver to stimulate ANS is head-up tilt (HUT). Tilt causes pooling of blood toward lower body and reduces the venous return to the heart. These activation of ANS leads to an increase of heart rate and peripheral vascular resistance aiming to maintain arterial pressure near to the level preceding the challenge (baro-reflex control).

Methods: we study the effects of sympathetic stimulation on ANSS and ANSSi induced with two different tilt at 45 and 90 degrees angles. We compare the ANSS and ANSSi with HRV analysis and baro-reflex control analysis. We plan to study 7 volunteers to detect a difference of 30 (standard deviation of 15) between the mean of ANSS and ANSSi at baseline and during tilt, with a power of 80% and alfa error of 5%.

ELIGIBILITY:
Inclusion Criteria:

* adult healthy humans (american society of anesthesiologists class I)
* age between 25 and 35 years old
* no assumption of any drug, beverages containing caffeine or alcohol during the previous 24 hours
* fasting 3 hours before the study protocol

Exclusion Criteria:

* american society of anesthesiologists class >1
* age <25 or >35 years
* pregnancy
* accidental discover of non sinus cardiac rhythm or ectopic beats >5%

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2013-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
to measure the degree of correlation of ANSS and ANSSi with LF/HF and baroreflex sensitivity and their agreement in response to an orthostatic sympathetic load | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera "Luigi Sacco" - Polo Universitario - University of Milan, Milan, Italy

REFERENCES:
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Bonhomme V, Uutela K, Hans G, Maquoi I, Born JD, Brichant JF, Lamy M, Hans P. Comparison of the surgical Pleth Index with haemodynamic variables to assess nociception-anti-nociception balance during general anaesthesia. Br J Anaesth. 2011 Jan;106(1):101-11. doi: 10.1093/bja/aeq291. Epub 2010 Nov 4. PMID 21051493
- [Background] Hamunen K, Kontinen V, Hakala E, Talke P, Paloheimo M, Kalso E. Effect of pain on autonomic nervous system indices derived from photoplethysmography in healthy volunteers. Br J Anaesth. 2012 May;108(5):838-44. doi: 10.1093/bja/aes001. Epub 2012 Feb 26. PMID 22369767
- [Background] Paloheimo MP, Sahanne S, Uutela KH. Autonomic nervous system state: the effect of general anaesthesia and bilateral tonsillectomy after unilateral infiltration of lidocaine. Br J Anaesth. 2010 May;104(5):587-95. doi: 10.1093/bja/aeq065. Epub 2010 Mar 30. PMID 20354006
- [Background] Montano N, Ruscone TG, Porta A, Lombardi F, Pagani M, Malliani A. Power spectrum analysis of heart rate variability to assess the changes in sympathovagal balance during graded orthostatic tilt. Circulation. 1994 Oct;90(4):1826-31. doi: 10.1161/01.cir.90.4.1826. PMID 7923668
- [Background] Pagani M, Lombardi F, Guzzetti S, Rimoldi O, Furlan R, Pizzinelli P, Sandrone G, Malfatto G, Dell'Orto S, Piccaluga E, et al. Power spectral analysis of heart rate and arterial pressure variabilities as a marker of sympatho-vagal interaction in man and conscious dog. Circ Res. 1986 Aug;59(2):178-93. doi: 10.1161/01.res.59.2.178. PMID 2874900
- [Background] Cooke WH, Hoag JB, Crossman AA, Kuusela TA, Tahvanainen KU, Eckberg DL. Human responses to upright tilt: a window on central autonomic integration. J Physiol. 1999 Jun 1;517 ( Pt 2)(Pt 2):617-28. doi: 10.1111/j.1469-7793.1999.0617t.x. PMID 10332107
- [Background] Kamiya A, Iwase S, Sugiyama Y, Mano T, Sudoh M. Vasomotor sympathetic nerve activity in men during bed rest and on orthostasis after bed rest. Aviat Space Environ Med. 2000 Feb;71(2):142-9. PMID 10685588
- [Derived] Colombo R, Marchi A, Borghi B, Fossali T, Rech R, Castelli A, Corona A, Guzzetti S, Raimondi F. Pulse Photoplethysmographic Analysis Estimates the Sympathetic Activity Directed to Heart and Vessels. Anesthesiology. 2015 Aug;123(2):336-45. doi: 10.1097/ALN.0000000000000712. PMID 26035252